CLINICAL TRIAL: NCT06670755
Title: A Clinical Trial Evaluating the Safety of an Aerosol BCG Controlled Human Infection Model in Assessing the Immunogenicity of Historical BCG Vaccination and Vaccination With ID93/GLA-SE in Healthy Adult Volunteers
Brief Title: ID93/GLA-SE Vaccination + BCG Challenge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TB045
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: This is a phase 1b vaccine efficacy study of ID93/GLA-SE in historically BCG-vaccinated and BCG-naïve healthy adult volunteers using an aerosol BCG challenge model.
  There will be four study groups with twelve volunteers in each group. Volunteers will be randomized to eligible groups based upon their BCG vaccine status, and will either be given 2 μg ID93 + 5 μg GLA-SE at Day 0 and Day 56 (Group A and C) prior to BCG aerosol challenge, or proceed directly to BCG aerosol challenge without vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: 2 doses of ID93/GLA-SE with 1 x 10^6 cfu BCG (historically BCG-vaccinated group) (Experimental): 12 historically BCG-vaccinated volunteers will be vaccinated with 2 doses of ID93/GLA-SE and after 112 days receive 1 x 10^6 cfu aerosol inhaled BCG as a challenge. All Group A volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: ID93/GLA-SE; Biological: BCG Danish
- Group B: 1 x 10^6 cfu BCG (historically BCG-vaccinated group) (Experimental): 12 historically BCG-vaccinated volunteers will receive 1 x 10^6 cfu aerosol inhaled BCG. All Group B volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish
- Group C: 2 doses of ID93/GLA-SE with 1 x 10^6 cfu BCG (BCG-naïve group) (Experimental): 12 BCG-naïve volunteers will be vaccinated with 2 doses of ID93/GLA-SE and after 112 days receive 1 x 10^6 cfu aerosol inhaled BCG as a challenge. All Group C volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: ID93/GLA-SE; Biological: BCG Danish
- Group D: 1 x 10^6 cfu BCG (BCG-naïve group) (Experimental): 12 BCG-naïve volunteers will receive 1 x 10^6 cfu aerosol inhaled BCG. All Group D volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish

INTERVENTIONS:
Biological: ID93/GLA-SE — ID93/GLA-SE is a protein-adjuvant vaccine which has been purposefully designed to elicit a diverse immune response against M.tb bacterial antigens, improve treatment outcomes and prevent TB disease in people already infected with M.tb.
  ID93/GLA-SE will be administered intramuscularly.
  Arms: Group A: 2 doses of ID93/GLA-SE with 1 x 10^6 cfu BCG (historically BCG-vaccinated group); Group C: 2 doses of ID93/GLA-SE with 1 x 10^6 cfu BCG (BCG-naïve group)
Biological: BCG Danish — BCG Danish 1331 is on the WHO list of pre-qualified vaccines and has a well-defined side effect profile. BCG is licensed for delivery via the intradermal route. It is not licensed for delivery via the aerosol route.
  For the challenge, aerosol BCG will be administered via nebulizer.

SUMMARY:
The purpose of this study is to:

1. Demonstrate the safety of a novel TB vaccine (ID93/GLA-SE) when given to both BCG-vaccinated and BCG-naïve volunteers.
2. Provide preliminary immunogenicity data of this novel TB vaccine (ID93/GLA-SE).

This clinical trial will apply an aerosol BCG challenge model involving 48 participants - 24 historically BCG-vaccinated volunteers and 24 BCG-naïve volunteers. Bronchoscopies will be performed 14 days post-challenge to measure BCG recovered from bronchial samples. Blood tests will be taken to look at potential immunological markers of immunity.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the deadliest infectious diseases worldwide. Key research priorities include the development of an effective vaccine.

Currently, the only licensed vaccine against TB is BCG (Bacille Calmette-Guérin). This works well against TB in childhood but is often ineffective in adults. Developing a new TB vaccine is difficult, as it is hard to determine which will be effective. In other diseases, e.g. influenza or malaria, it is possible to experimentally-infect volunteers with the disease to see if the proposed vaccine is effective. This is called a "controlled human challenge or infection model" and is possible in easily treatable or self-limiting diseases. This is not possible with TB, where treatments may be harmful and complex. Using BCG, a live attenuated (weakened) strain of the bacteria that do not cause disease in healthy individuals, the investigators have developed a challenge model to mimic TB infection.

Mycobacterium tuberculosis, the bacterium that causes TB, infects people by inhalation into the lungs. Therefore, inhaled BCG more closely imitates TB infection than an injection. Previous studies (TB041 and TB043) and a current study (TB044) in our group used aerosol inhaled BCG in both previously BCG-vaccinated and BCG-naïve volunteers to show that aerosolised BCG could be safely employed, and that BCG could be detected in lung washings two weeks after challenge.

A novel TB vaccine (ID93/GLA-SE) has recently undergone clinical trials (phase IIa) to show that it can be given safely to healthy people. Its ability to protect people from TB is currently being investigated.

The purpose of this study is to show the safety of this approach and provide preliminary immunogenicity data of this novel TB vaccine (ID93/GLA-SE) in both historically BCG-vaccinated and BCG-naïve volunteers, using an aerosol BCG challenge model. It will involve 48 participants; 12 historically BCG-vaccinated and 12 BCG-naïve participants will initially receive 2 injections of the intramuscular ID93/GLA-SE before challenge with aerosol BCG, while a further 24 participants (12 historically BCG vaccinated) will have aerosol BCG challenge alone. Bronchoscopies will be performed 14 days post aerosol BCG challenge to measure BCG recovered from bronchial samples. Blood samples will be taken to look at potential immunological markers of protection.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18-55 years
* Resident in or near Oxford for the duration of the study period
* Provide written informed consent
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner (or review summary care record, if available)
* Allow the investigator to register volunteer details with a confidential database (The Over-volunteering Protection Service) to prevent concurrent entry into clinical studies/trials
* Agreement to refrain from blood donation during the course of the study
* For persons of child-bearing potential only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening, vaccination, challenge and bronchoscopy
* Able and willing (in the investigator's opinion) to comply with all study requirements
* No clinically relevant findings in medical history or on physical examination
* Screening IGRA (interferon gamma release assay) negative
* Willing to be tested for evidence of COVID-19 infection and to allow public health notification of the results if required
* EITHER Previously vaccinated with the BCG (at least 12 months prior to enrolment, as evidenced by a visible scar or documentation in medical or occupational health records) OR Never previously vaccinated with BCG and no evidence of BCG scar at physical examination

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment or during the trial follow up period
* Any clinically significant respiratory disease, including asthma
* Current smoker (defined as any smoking including e-cigarettes in the last 3 months)
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study agent, any essential study procedure, sedative drugs, or any local or general anaesthetic agents
* History of allergic reaction to Kanamycin or kanamycin-related antibiotics
* Clinically significant history of skin disorder, allergy, atopy, cancer (except basal cell carcinoma of the skin or carcinoma in situ of the cervix), bleeding disorder, cardiovascular disease (including uncontrolled hypertension), gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* Any significant autoimmune conditions or immunodeficiency (including current HIV)
* Previous diagnosis or treatment for TB disease or latent TB infections
* Clinical, radiological, or laboratory evidence of current active TB disease or latent TB infection
* Previous receipt of any investigational TB vaccine or aerosolised BCG
* Currently infected with HIV, Hepatitis B or Hepatitis C based on positive serological testing (Hepatitis B surface antigen, Hepatitis C virus or HIV antibodies) and confirmatory molecular testing if indicated
* Concurrent use of oral, inhaled or systemic steroid medication or use for more than 14 days within the last 6 months (steroids used as a cream or ointment are permissible), or the use of other immunosuppressive agents concurrently or for more than 14 days within the last 6 months
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned enrolment date
* Administration of a live vaccine within the preceding 28 days prior to enrolment, or plan for such prior to aerosol challenge
* Administration of any other non-live vaccine within the preceding 14 days prior to enrolment
* Current use of any medication or other drug taken through the nasal or inhaled route including cocaine or other recreational drugs
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Pregnancy, lactation or intention to become pregnant during study period
* Previously resident for more than 12 months concurrently in the rural areas of a tropical climate where significant non-tuberculous mycobacterial exposure is likely
* Shares a household with someone with clinically significant immunodeficiency (either from infection or medication) who is deemed to be at risk of developing disseminated BCG infection if exposed to BCG
* Clinically significant abnormality on screening chest radiograph
* Clinically significant abnormality of lung function testing
* Any clinically significant abnormality of screening blood or urine tests
* A body mass index (BMI) of <18.5 or >45
* Any other significant disease, disorder, or finding, which, in the opinion of the investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety of BCG challenge by the aerosol inhaled route in healthy volunteers and recently ID93/GLA-SE-vaccinated adult volunteers. | Group A and C - up to day 168, Group B and D - up to day 56 (Adverse events are collected throughout the duration of the study. Specific timepoints for blood and lung function tests have been mentioned in the measure description.)
  Safety will be assessed through actively and passively collected data on adverse events, detailed participant symptom profiles, and lung function test results.
  Adverse events will be collected at each visit and via diary card. Safety blood tests will be performed at baseline, day 14 and day 70. Lung function tests will be performed at day 0 post challenge and day 28, as well as later time points if clinically indicated.

SECONDARY OUTCOMES:
Differences in colony forming units recoverable of ID93/GLA-SE against a controlled human aerosol BCG infection model. | On day 14 post-challenge
  Difference in BCG recovery from bronchoalveolar lavage fluid 2 weeks after BCG aerosol challenge between ID93/GLA-SE and naïve arms, investigated using time to positivity (number of hours or days for the BCG to flag in the mycobacterium growth indicator tube (MGIT)) and mycobacterial speciation.
  Bronchoscopies will be performed 14 days post-challenge. Respiratory samples will be cultured for BCG.

OTHER OUTCOMES:
Exploratory outcome: Immunological and microbiological markers that correlate with the levels of BCG recovered from bronchial and other samples after vaccination with ID93/GLA-SE in BCG-naïve and historically BCG-vaccinated volunteers. | Group A and C - up to day 168, Group B and D - up to day 56.
  Further exploratory research will be performed on blood and respiratory samples collected on the volunteers throughout the study. Examples of research that may be performed include: ex-vivo ELISpot and ELISAs on blood samples, RNA sequence analysis and intracellular cytokine staining of blood, molecular diagnostics on blood or bronchial samples.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Professor, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom